CLINICAL TRIAL: NCT03772769
Title: Diagnostic Modalities for Severe Odontogenic Infections Using Rapid, Target Enriched Multiplex PCR (TEM- PCR)
Brief Title: Diagnostic Modalities for Severe Odontogenic Infections Using Rapid, Target Enriched Multiplex PCR (TEM- PCR) by Diatherix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Eurofins (Industry)
Responsible Party: Principal Investigator, Nagi Demian, Clinical Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-DB-18-0506
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Odontogenic Deep Space Neck Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with advanced deep space odontogenic infection (Experimental): Subjects will be diagnosed via two methods: 1. Target Enriched Multiplex PCR (TEM- PCR) and 2. Standard microbial culture.
  Interventions: Diagnostic Test: Target Enriched Multiplex PCR (TEM- PCR); Diagnostic Test: Microbial culture

INTERVENTIONS:
Diagnostic Test: Target Enriched Multiplex PCR (TEM- PCR) — Target Enriched Multiplex PCR (TEM- PCR) assays will be performed and will probe for the typical array of advanced deep space odontogenic infections, as well as MRSA resistance, clindamycin resistance, and the presence of Panton-Valentine leukocidin (PVL) toxin, a toxin produced by some bacteria.
Diagnostic Test: Microbial culture — Standard diagnosis by microbial culture.

SUMMARY:
The purpose of the study is to evaluate the sensitivity and specificity of the Target Enriched Multiplex (TEM) polymerase chain reaction (PCR) platform for the rapid molecular diagnosis and treatment of odontogenic deep space neck infections.

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom there is clinical and radiographic evidence of an odontogenic deep space neck infection.

Exclusion Criteria:

* Patients with gross communication between the abscess and the oral cavity will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Specificity as assessed by number of participants who had matching results between TEM-PCR and standard microbial culture | Baseline (at the time the sample was obtained from the patient)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Jundt, DDS, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Th University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No